CLINICAL TRIAL: NCT03854422
Title: Which Position is Suitable for Easy, Fast and Comfortable Colonoscopy
Brief Title: For Easy, Fast and Comfortable Colonoscopy, Which Position
Acronym: EFC_COLON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, BETÜL TOPAL, research assistant doctor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EasyCOLON study
Record Dates: First submitted 2019-01-11; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Colonic Diseases, Functional; Prone Position; Endoscopy
Keywords: Colonoscopy; Insertıon tecnique; Prone; Left Supine; Dynamic
MeSH Terms: conditions — Colonic Diseases, Functional | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: this study includes 3 different groups. left, left supine,dynamıc
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Left Position during colonoscopy (Active Comparator): Left position, the patient will be in the left-side position during the entire colonoscopy period. If necessary, change of position and pressure will be allowed. During this procedure, the time to reach the cecum and terminal ileum, patient comfort, and the process memory lost will be measured.Moreover, process recall, sedation amounts and pain scale will be measured after the procedure..During the process, it will be examined whether there is any need for loop formation, repositioning requirement and pressure requirements. The type and amount of anesthetic agent (midazolam) used during the process is paid attention to be equal. All procedures will be done with the same brand device. After the procedure, a mini questionnaire will be applied to the patients for the pain scale.
  Interventions: Device: left position
- Left Supine Position during colonoscopy (Active Comparator): Left Supine position, the patient will be in the left and supine ( after splenic flexura) position during the entire colonoscopy period. If necessary, change of position and pressure will be allowed. During this procedure, the time to reach the cecum and terminal ileum, patient comfort, and the process memory lost will be measured.
  Interventions: Device: left supine position
- Dynamic position during colonoscopy (Active Comparator): Dynamic position, the patient will be stared as left position during colonoscopy period. If necessary, change of position and pressure will be allowed at any time. During this procedure, the time to reach the cecum and terminal ileum, patient comfort, and the process memory lost will be measured..During the process, it will be examined whether there is any need for loop formation, repositioning requirement and pressure requirements. The type and amount of anesthetic agent used during the process is paid attention to be equal. The use of midazolam as an anesthetic agent was planned.All procedures will be done with the same brand device. After the procedure, a mini questionnaire will be applied to the patients for the pain scale.
  Interventions: Device: dynamic position

INTERVENTIONS:
Device: left position — colonoscopy will be performed in 3 different locations. Left position, the patient will be in the left-side position during the entire colonoscopy
  Other Names: Colonoscopy in the Left position
  Arms: Left Position during colonoscopy
Device: left supine position — Colonoscopy in the Left supine position
  Arms: Left Supine Position during colonoscopy
Device: dynamic position — Colonoscopy in the Dynamic position
  Arms: Dynamic position during colonoscopy

SUMMARY:
Colonoscopy is one of the most common endoscopic procedures today. However, it sometimes can be a serious challenging situation both for the clinicians and patients. In this study, the investigators tried to determine which colonoscopic position allows easy, fast and comfortable way.

DETAILED DESCRIPTION:
colonoscopy and colonoscopic screening are the most common routine studies to reduce the incidence of colorectal cancer.In this process, the most important problem for the endoscopist and the patient is pain, loop formation, (the reason why the device is not able to progress in the bowel) and in some patients it takes a long time due to these reasons and the risk of complication development.The subject of what should be the most ideal position in colonoscopy has previously been studied in some specific subgroups.There is not enough study on what should be the ideal position in colonoscopy. In this study, the investigators tried to determine which colonoscopic position allows easy, fast and comfortable way.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged for 18 to 80 years,
* colonoscopy indications (iron deficiency anemia ,Malignancy screening in patients over 50 years of age,secret blood positivity in stool, rectal bleeding,patients describing Hematoconia, chronic diarrhea, constıpatıon

Exclusion Criteria:

* patients with previous colon surgery
* serious comorbid disease (congestive heart failure ef< %30 , advanced chronic obstructive pulmonary disease,terminal period cancer with a life expectancy of less than 5 years, those who have not had appropriate bowel cleaning,endoscopic treatment during colonoscopy or removal of diagnostic lesions,other sedatives for sedation other than midazolam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
Time to reach cecum | 2 hour
  Cecum intubation time is the insertion time taken from first visualization of rectal mucosa to cecum

SECONDARY OUTCOMES:
patient's comfort assessment: Visual Analog Score | 3 hour
  patients' discomfort will be assessed by a 10-cm visual analog scale, in which a score of 0 denoted no pain and a score of 10 denoted unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: TARIK AKAR, MD, Study Director — BULENT ECEVIT UNIVERSITY FACULTY OF MEDICINE , GASTROENTEROLOGY
Locations (1):
- Betul Topal, Zonguldak, Kozlu Bulent Ecevit University Faculty of Medicine, Turkey (Türkiye)